CLINICAL TRIAL: NCT04054206
Title: Relative Bioavailability Study of an Extended Release (ER) Tablet Formulation of MN-166 (Ibudilast) Compared to an Intermediate Release (IR) Capsule Formulation in Healthy Volunteers
Brief Title: Relative Bioavailability of MN-166 (Ibudilast) in Extended Release Tablet vs. Intermediate-release Capsule in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: MediciNova (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: MN-166-HDT-002
Record Dates: First submitted 2019-08-06; First posted 2019-08-13 (Actual); Last update posted 2020-07-15 (Actual); Status verified 2020-07

CONDITIONS: Healthy Volunteers
MeSH Terms: interventions — ibudilast

STUDY DESIGN:
Intervention Model Description: 12 healthy male and female participants (enrollment is 6 female and 6 male participants). Each enrolled/consented participant will be randomly assigned to 1 of 6 treatment sequences which consists of 3 treatments (ER fasted, ER fed, and IR fasted) in a crossover design, administered one week apart.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Sequence 1 (Active Comparator): Two participants will be randomly assigned to sequence 1 comprising 3 treatments (ER fasted, ER fed, and IR fasted) in a crossover design, administered one week apart:
  Day 1-7: ER fasted; Day 8-15: ER fed Day 15-22: IR fasted
  Interventions: Drug: MN-166
- Sequence 2 (Active Comparator): Two participants will be randomly assigned to sequence 2 comprising 3 treatments in a crossover design, administered one week apart: Day 1-7: ER fed; Day 8-15: IR fasted; Day 15-22: ER fasted
  Interventions: Drug: MN-166
- Sequence 3 (Active Comparator): Two participants will be randomly assigned to sequence 3 comprising 3 treatments in a crossover design, administered one week apart:
  Day 1-7: IR fasted; Day 8-15: ER fasted; Day 15-22: ER fed
  Interventions: Drug: MN-166
- Sequence 4 (Active Comparator): Two participants will be randomly assigned to sequence 4 comprising 3 treatments in a crossover design, administered one week apart:
  Day 1-7: IR fasted; Day 8-15: ER fed; Day 15-22: ER fasted
  Interventions: Drug: MN-166
- Sequence 5 (Active Comparator): Two participants will be randomly assigned to sequence 5 comprising 3 treatments in a crossover design, administered one week apart:
  Day 1-7: ER fasted; Day 8-15: IR fasted; Day 15-22: ER fed
  Interventions: Drug: MN-166
- Sequence 6 (Active Comparator): Two participants will be randomly assigned to sequence 6 comprising 3 treatments in a crossover design, administered one week apart:
  Day 1-7: ER fed; Day 8-15: ER fasted; Day 15-22: IR fasted
  Interventions: Drug: MN-166

INTERVENTIONS:
Drug: MN-166 — MN-166 (ibudilast) is an orally available small molecule drug currently being investigated for human treatment in multiple sclerosis, amyotrophic lateral sclerosis, glioblastoma, and alcohol and drug use disorders.
  Other Names: ibudilast; Pinatos capsule

SUMMARY:
This study will investigate the PK, relative bioavailability, safety, and tolerability of the extended release (ER) 50 mg MN-166 (ibudilast) tablet formulation as compared to the intermediate-release (IR) capsule formulation of MN-166 (ibudilast) and to examine the effect of food on the pharmacokinetics of the ER formulation.

DETAILED DESCRIPTION:
This is a Phase 1, open-label, single-center study in at least 12 healthy volunteers or participants.

Participants (at least n=2/sequence) meeting study eligibility and providing informed consent will be randomized to one of six treatment sequences. The three treatments of each sequence will be administered in a crossover fashion, separated by one week apart. Thus, participation in the study is 3 weeks long per participant.

During each single-dose treatment, participants will check in the study facility the night before dosing and remain at the facility until 32 hours after dosing. For example, the participant would arrive at the study facility at 8:00 PM Sunday night, receive a single dose at 8:00 AM Monday morning, and blood samples will be taken prior to dosing and 30 minutes, 1, 2 4, 6, 8, 10, 12, 24, and 32 hours after dosing. After the 32-hour sample collection, participants may leave the study facility. Participants will return to the study facility for outpatient visits at each remaining PK sampling day (48, 72, and 96 hours after dosing) and after last treatment in each sequence. Participants will be discharged from the study after the last treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Able to provide written informed consent.
2. Healthy non-smoking male and female subjects aged 18 to 45 years, inclusive. Health status is determined by physical examination, medical history, no clinical abnormalities in laboratory and urine analyses, normal renal function, liver enzymes less than twice the upper limit of normal (ULN), and electrocardiogram (ECG) with QT interval adjusted for heart rate within normal limits at the screening visit.
3. A body mass index (BMI) of 18 kg/m2 or greater, but less than 36 kg/m2.
4. Agree to use barrier contraceptive methods during the course of the study (hormonal contraceptive alone is not acceptable).
5. Females of child-bearing potential must have a negative urine pregnancy test on Day 1. If post-menopausal female, follicle stimulating hormone (FSH) level > 40 IU/L.

Exclusion Criteria:

1. History of clinically significant drug allergy or anaphylaxis, including known hypersensitivity to Pinatos® or its components.
2. History of any condition(s) which might affect drug absorption, metabolism or excretion.
3. Clinical evidence or a history of clinically significant cardiovascular, respiratory, renal, hepatic, gastrointestinal, hematological, neurologic, or other chronic disease as judged by the Investigator.
4. History of severe psychiatric disease, especially major depression. Severe psychiatric disease is defined as treatment with an antidepressant medication or a major tranquilizer at therapeutic doses for major depression or psychosis, respectively, for at least 3 months at any previous time or any history of the following: a suicidal attempt, hospitalization for psychiatric disease, or a period of disability due to a psychiatric disease.
5. History of severe cardiac disease [e.g., New York Heart Association (NYHA) Functional Class III or IV], myocardial infarction within 6 months, ventricular tachyarrhythmias requiring ongoing treatment, unstable angina or other significant cardiovascular diseases.
6. Estimated creatinine clearance outside the normal range (</= 80 mL/min) at screening.
7. History or other evidence of severe illness or any other conditions which would make the subject, in the opinion of the investigator, unsuitable for the study.
8. Evidence of alcohol and/or drug abuse within one year of screening.
9. Positive results on screen for drugs of abuse or alcohol at screening visit or Day 0.
10. History within 1 year of screening visit, or current habit, of smoking more than 10 cigarettes per day or equivalent (>3 cigars or >3 pipes-full).
11. Donated blood in the past 90 days or have poor peripheral venous access.
12. Platelets < 100,000/mm3, history of thrombocytopenia.
13. Confirmed diagnosis of chronic liver disease, for example, chronic Hepatitis B, Hepatitis C infection, auto-immune, alcoholic or neoplastic liver disease.
14. Positive serostatus for HIV, HCV, or HBV.
15. Currently pregnant or nursing.
16. Male partners of females who are pregnant.
17. History of clinically significant cardiovascular, pulmonary, endocrine, neurological, metabolic, or psychiatric disease.
18. Participation in a clinical study with an investigational drug, biologic, or device within 3 months before receiving study drug.
19. Used any systemic medications, including vitamins and over-the-counter items, during the 14 days (or five times the elimination half-life of the medication, whichever is longer) before receiving study drug or will require their use during the study. Metabolic inducers and herbal preparations, which have been shown to produce metabolic enzyme induction or inhibition, whether as teas or formulations, are prohibited 28 days before dosing. Paracetamol 3000 mg/day will be allowed up to 2 consecutive days before dosing and during the outpatient phase of the study, as needed.
20. Unable to swallow large tablets.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2019-06-24 (Actual); Primary Completion 2019-07-17 (Actual); Study Completion 2020-05-31 (Actual)

PRIMARY OUTCOMES:
Compare the pharmacokinetic profile of ER and IR formulations in single-dose administration of MN-166 (ibudilast) | From the time of pre-dose (immediately prior to taking the assigned MN-166/ibudilast formulation) to 0.5, 1, 2, 4, 6, 8, 10, 12, 24, 32, 48, 72, 96, and 168 hours post-single treatment dose.
  Compare the maximum plasma concentrations (Cmax) of MN-166 (ibudilast) of ER 50 mg tablet and IR 10 mg capsule (5 capsules) formulations, in a single-dose regimen in healthy volunteers.
Compare the pharmacokinetic profile of ER and IR formulations in single-dose administration of MN-166 (ibudilast) under fed or fasting states | From the time of pre-dose (immediately prior to taking the assigned MN-166/ibudilast formulation under either feeding or fasting conditions) to 0.5, 1, 2, 4, 6, 8, 10, 12, 24, 32, 48, 72, 96, and 168 hours post-single treatment dose.
  Cmax of MN-166 (ibudilast) of ER 50 mg tablet and IR 10 mg capsule (5 capsules) formulations, in a single-dose regimen in healthy volunteers fed a high-fat meal 1 hour prior to dosing or fasted 8 hours prior to dosing.

SECONDARY OUTCOMES:
Number of healthy volunteers with treatment-related adverse events as assessed by CTCAE v.4.0 | From the time of pre-dose (immediately prior to taking the assigned MN-166/ibudilast formulation under either feeding or fasting conditions) to 0.5, 1, 2, 4, 6, 8, 10, 12, 24, 32, 48, 72, 96, and 168 hours post-single treatment dose.
  Compare the number and frequency of treatment-emergent adverse events (serious and non-serious) profiles of ER and IR formulations of MN-166 (ibudilast) in healthy volunteers.
Changes in physical exam results | From the night before single-dose treatment to 168 hours post-dose under fed and fasted conditions.
  Compare the number and frequency of clinically significant changes in physical exam results between ER and IR formulations of MN-166 (ibudilast) in healthy volunteers.The HV's general health (for example, appearance, presence of illness or injury; temperature, pulse, or heart rate indicative of a concurrent illness) will be assessed to determine whether or not to continue in the study.
Number of participants with clinically significant abnormal laboratory results | From the night before single-dose treatment to 168 hours post-dose under fed and fasted conditions.
  Compare the frequency of clinically significant abnormal laboratory results of ER and IR formulations of MN-166 (ibudilast) in healthy volunteers under fed and fasted states.

CONTACTS AND LOCATIONS:
Overall Officials: David P Walling, PhD, Principal Investigator — Collaborative Neuroscience Network, LLC
Locations (1):
- Collaborative Neuroscience Network, Garden Grove, California, United States